CLINICAL TRIAL: NCT05233319
Title: A Single-Center, Prospective Clinical Study to Demonstrate That mCVI(R) Accurately Captures Pulse Rate and Respiratory Rate in 20 Healthy Volunteers in Comparison to Traditional Measurements of the Nonin Lifesense Capnograph
Brief Title: mCVI Confirmatory Clinical Study: Algorithm Verification With Healthy Volunteers
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding, project not being pursued
Sponsor: Intelomed, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mCVI004
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Algorithm Verification

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
This single center confirmatory clinical study is to verify the algorithm of mCVI® to accurately capture pulse rate and respiratory rate in 20 healthy subjects in comparison to traditional measurements of the Nonin Lifesense Capnograph. This is a non significant risk device.

DETAILED DESCRIPTION:
In this confirmatory clinical study the mCVI® device is a mobile application used to simply verify the algorithm when the mobile video reads a patients pulse rate and respiratory rate while spontaneously breathing. There is no facial recognition technology. There is no immediate feedback given to the research team to act upon or provide for further clinical care decisions. In real time, the mCVI® device will be compared to traditional measurements of the Nonin Lifesense Capnograph.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 21 - 70

Exclusion Criteria:

* Medical conditions that could compromise a participant's ability to provide for all breathing samples, pedal the Cubii Pro elliptical, or follow instructions
* Medications that could compromise a participant's ability to participate in the study
* Documented medical history of respiratory or cardiovascular disease
* Excessive facial hair, facial deformities, or obstructions (like glasses or face masks/shields) that could compromise the recording of pulse rate and respiratory rate of the mCVI®
* Any face lotions or make up foundations that could compromise the recording of pulse rate and respiration rate of the mCVI®
* Recent (≤ 1 month) surgical procedure of any kind
* Current participation in another investigational clinical trial
* Inability to provide informed consent

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pulse Rate Verification | 1 month
  To demonstrate that mCVI(R) accurately captures pulse rate comparison to Nonin Lifesense Capnograph
Respiration Rate Verification | 1 month
  To demonstrate that mCVI(R) accurately captures respiratory rate in comparison to Nonin Lifesense Capnograph

SECONDARY OUTCOMES:
Skin Tone Pulse Rate Verification | 1 month
  To demonstrate that mCVI(R) accurately captures pulse rate in healthy volunteers with a variety of skin tones
Skin Tone Respiration Rate Verification | 1 month
  To demonstrate that mCVI(R) accurately captures respiration rate in healthy volunteers with a variety of skin tones

CONTACTS AND LOCATIONS:
Locations (1):
- InteloMed, Inc., Cranberry Township, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No